CLINICAL TRIAL: NCT02642835
Title: A Long Term Follow up of Perigee Anterior Meshes Performed for Recurrent Prolapse
Brief Title: A Long Term Follow up of Anterior Meshes for Recurrent Prolapse
Status: Completed | Type: Observational
Sponsor: Medway NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Professor Jonathan Duckett, Consultant Urogynaecologist, Medway NHS Foundation Trust
Other Study IDs: 9/12/14
Record Dates: First submitted 2015-08-27; First posted 2015-12-30 (Estimated); Results first posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2016-03

CONDITIONS: Genital Diseases, Female; Pelvic Organ Prolapse
Keywords: mesh; pelvic organ prolapse
MeSH Terms: conditions — Genital Diseases, Female; Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: vaginal wall mesh — retrospective review of case series

SUMMARY:
Prolapse of the vaginal wall and uterus are common conditions affecting up to 50% of parous women. The socioeconomic, psychological and physical impacts of prolapse are considerable. 11% of women will undergo a surgical repair by the age of 80 years. The commonest compartment affected is the anterior vaginal wall. Unfortunately there is a significant rate of recurrent prolapse or a failure of the primary procedure. This has lead to the introduction of new techniques and the use of different materials to augment the repair. Mesh augmented repairs aim to reduce the rate of recurrent prolapse. However, the use of synthetic mesh is associated with complications which are not found in non mesh repairs. 10% of women will have a mesh complication of which 70% will require a further surgical procedure to manage the complication. There are extra costs associated with purchasing the mesh, with longer operating times to insert the mesh and managing complications caused by the mesh. Balancing the extra risks of mesh surgery against the benefits is probably one of the most contentious issues in urogynaecology at the present time.

Regulatory authorities in the USA (FDA) and UK (MHRA) have become increasingly interested in the use of mesh to support the vaginal wall in prolapse surgery due to risks and complications being reported. To date there is little evidence regarding the long term safety and efficacy of anterior mesh repairs. This study aims to rectify this deficiency for Perigee.

DETAILED DESCRIPTION:
This will be a consecutive cohort study of patients identified from a surgical database of Perigees performed in a single centre. All patients will have had the procedure performed between 2007 and 2011. This will be a single centre study. The principle investigator has both electronic and hand written records of all Perigee repairs performed since the introduction of this technique in 2007. The patients will be identified from both the paper and electronic databases and cross referenced.

After obtained appropriate ethical approval, patients identified as having a perigee mesh inserted will be asked to attend Medway Hospital for a full clinical evaluation. They will be sent a letter with an appointment to come to the hospital. They will be asked to complete the Pelvic floor distress inventory questionnaire to assess their symptoms. They will have a pelvic examination to determine if they have any mesh erosion and will undergo a POP-Q score. This visit will take 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing a perigee procedure after January 2007

Exclusion Criteria:

* Patient having non mesh repairs over the same time scale

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients having previously undergone a mesh repair
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2015-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Duckett, FRCOG, Principal Investigator — Medway NHS Foundation Trust
Locations (1):
- Medway NHS Foundation trust, Gillingham, Kent, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Mesh Group: all had an anterior mesh for recurrent prolapse
Period: Overall Study
Arm/Group | Mesh Group
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Mesh Group: underwent anterior mesh for recurrent cystocele
Arm/Group | Mesh Group
Number analyzed (Participants) | 48
Age, Continuous [Mean (Full Range); unit: years] | 66 [47 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 0
BMI [Mean (Full Range); unit: wt kg/ht m squared] | 27.4 [19 to 44]
Parity [Median (Full Range); unit: vaginal deliveries past 28 weeks] | 2 [1 to 4]
time to follow up (months) [Mean (Full Range); unit: number of months] | 82 [48 to 106]

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With a Current Mesh Erosion or Treated for a Mesh Erosion Since Inserted
Description: clinic visit. 5 patients were interviewed by phone and were not examined - hence this figure is out of 43 not 48.
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Mesh Group
Number analyzed (Participants) | 43
Participants | 5

2. Secondary Outcome: Number of Participants With no Physical Evidence of Recurrent Prolapse as Determined by Physical Examination
Description: The presence of less than stage 2 prolapse (eg stage 1) anterior wall prolapse determined as anatomical success. A stage one prolapse is higher than 1cm above the vaginal entrance.
  A stage 2 prolapse means that the leading edge of the prolapse is between 1cm above the entrance to the vagina up to 1cm below the entrance to the vagina.
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Mesh Group
Number analyzed (Participants) | 43
Participants | 26

3. Secondary Outcome: Number of Participants Complaining of a Bulge. Recurrent Prolapse
Description: Efficacy determined by the question in the pelvic floor prolapse distress inventory "usually have a bulge or something falling out that you can see or feel in your vaginal area". Determined at clinic visit by questioning
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Mesh Group
Number analyzed (Participants) | 48
Participants | 14

4. Secondary Outcome: Number of Participants Requiring Treatment for Recurrent Prolapse - Prolapse in the Same Part of the Vagina
Description: clinic visit; number of participants who underwent reoperation of recurrent prolapse in the same compartment
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Mesh Group
Number analyzed (Participants) | 48
Participants | 1

5. Secondary Outcome: Number of Participants Who Underwent Reoperation for Prolapse in a Different Compartment
Description: This is where the mesh has held up and there is no prolapse where it was inserted. This measure refers to when a different part of the vagina has prolapsed.
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Mesh Group
Number analyzed (Participants) | 48
Participants | 8

6. Secondary Outcome: Number of Participants Who Developed New Stress Incontinence
Description: The mesh has caused the prolapse to be successfully repaired but the patient has developed stress incontinence as a separate issue. clinic visit
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Mesh Group
Number analyzed (Participants) | 48
Participants | 5

7. Secondary Outcome: Number of Participants Who Rated Their Improvement as Better or Very Much Better
Description: The patient global impression of Improvement scale (PGI-I) is a global improvement scale filled out by the patient. It is graded as very much better, much better, a little better. no change, a little worse, much worse or very much worse.clinic visit
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Mesh Group
Number analyzed (Participants) | 48
Participants | 33

8. Secondary Outcome: Number of Participants Who Needed Surgical Mesh Removal for Erosion
Description: A mesh erosion is when the body rejects the mesh and it is visible in the vagina rather than being buried under the vaginal epithelium. clinic visit
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Mesh Group
Number analyzed (Participants) | 48
Participants | 2

9. Secondary Outcome: Number of Participants Who Needed Reoperations for Pain
Description: patients may develop pain after the original operation which needs a second surgical procedure to try and help. clinic visit
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Mesh Group
Number analyzed (Participants) | 48
Participants | 3

10. Secondary Outcome: Number of Participants Who Experienced Intraoperative Complications
Description: This records any problems that were encountered at the original insertion of the mesh. clinic visit
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Mesh Group
Number analyzed (Participants) | 48
Participants | 0

ADVERSE EVENTS:
Arm/Group | Mesh Group
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No